CLINICAL TRIAL: NCT05610371
Title: Intrauterine Anesthesia in Operative, Awake, Office Hysteroscopy. A Randomized Double-blind Placebo-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0054-19-AAA
Record Dates: First submitted 2022-10-23; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-09

CONDITIONS: Anesthesia, Local; Office Hysteroscopy
Keywords: hysteroscopy; lidocaine; see and treat
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: RCT double blind
Who Masked: Participant, Care Provider, Investigator
Masking Description: RCT double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine The study group (Experimental): The study group underwent hysteroscopy using saline to which 10ml of 2% lidocaine was added to the first 1000 ml.
  Interventions: Drug: Lidocaine; Drug: Saline
- Saline The control group (Placebo Comparator): The control group underwent hysteroscopy using a saline distension medium.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — The study group underwent hysteroscopy using saline to which 10ml of 2% lidocaine was added to the first 1000 ml. This dose of lidocaine was calculated to allow maximal benefits with minimal potential complications. The maximal dose of lidocaine is 5mg\kg in adults which translates to 200mg in a 40kg patient. We have set 200 mg as the maximal dose of lidocaine in our study, assuring the dosage is safe. The rest of the procedure following the first 1000ml of saline was completed using saline alone as needed.
  Other Names: Essracaine
  Arms: Lidocaine The study group
Drug: Saline — The control group underwent hysteroscopy using a saline distension medium.
  Other Names: Sodium chloride

SUMMARY:
Objective: to evaluate intrauterine lidocaine infusion effectiveness in reducing pain associated with operative, awake office hysteroscopy Methods: A total of 100 patients will be randomized for this study The control group underwent hysteroscopy using a saline distension medium. The study group underwent hysteroscopy using 10ml of 2% lidocaine that was added to the first liter of distension medium. Patients quantified their pain using a 0-10 VAS score, at the following five predefined points: baseline, before the procedure; while inserting the hysteroscope through the cervix; during the operative procedure; immediately after the procedure and 15 minutes following the procedure.

DETAILED DESCRIPTION:
1. Background

   Ambulatory hysteroscopy is a safe, feasible, and accurate procedure for diagnosing and treating intrauterine pathology. [1]

   Office hysteroscopy does not require hospital admission, preparatory tests, and general anesthesia. Importantly, it has decreased postsurgical recovery period, global cost of the procedure, and rate of complications. [2] New approaches have evolved due to technological advances in instrumentation, an office hysteroscopy that combines diagnosis and treatment of the pathology into a single clinical procedure is referred to as "See and Treat hysteroscopy" (SATH) [3].

   SATH allows diagnosis of different conditions affecting the uterine cavity in an office setting, followed immediately with treatment to resolve them, thus avoiding the patient having to undergo a subsequent procedure [4].

   Pain during or after the procedure can discourage patients from undergoing office diagnostic hysteroscopy or SATH. [5] and remains a significant cause for failure to complete the procedure.

   The type of anesthesia used depends on the procedure, the patient's level of anxiety, and the anesthesiologist's expertise. Simple diagnostic procedures can be performed without anesthesia, with a para-cervical block, or with mild sedation. In a meta-analysis reviewing 36 studies only para-cervical block demonstrated a significant anesthetic effect [Munro]. There is controversy about anesthesia and analgesia for outpatient hysteroscopy, as there is not enough high-quality evidence, and marked heterogeneity between trials makes it very difficult to draw generalizable conclusions.

   In a recent study we have evaluated the effect of distension medium composed of 0.9% saline solution with Lidocaine vs Saline alone and it's effect on pain in diagnostic hysteroscopy. No studies had been published regarding this method of analgesia in SATH, and it's effect on pain during the procedure and immediately following the procedure.
2. Aims

   The primary aim of the current study is to evaluate the effect of local instillation of lidocaine in relieving pain during office SATH hysteroscopy.

   Secondary aims include the rate of failure in performing the procedure and patient satisfaction among patients in the study group vs. controls.
3. Hypothesis

   In this prospective, randomized, double blind study, utilizing adult women undergoing office SATH hysteroscopy, local instillation of lidocaine in the distension media should reduce the pain during and following the procedure by 20% and also improve patient satisfaction and might reduce failure rates without an increase in complication rates.
4. Settings and participants

   All patients referred to a diagnostic office SATH hysteroscopy at the outpatient clinics in Assuta Ashdod University Hospital that fit the inclusion criteria.

   Inclusion criteria:

   • Women between the ages of 20 years - 52 years inclusive.

   • Undergoing SATH office hysteroscopy

   • Patients are able to provide written consent

   Exclusion criteria:

   • Previous Pelvic Inflammatory Disease (PID) or documented tubal occlusion
   * Inability to consent due to cognitive or language barrier
   * Allergy to Lidocaine
   * Documented failed hysteroscopy prior to the current referral
5. Study methodology and techniques

Study Design

This study is a prospective randomized double blind trial.

Women undergoing SATH office hysteroscopy that are eligible for the study will be divided into 2 groups:

1. Hysteroscopy using saline alone as a distension medium
2. Hysteroscopy using a 10 ml of 2% lidocaine in a 1000 ml of saline as a distension medium The distension medium bags will be prepared by the Assuta Ashdod University Hospital Pharmacy. The first bag will contain 10 ml of 2% lidocaine in a 1000 ml of saline or saline alone and will be coded using a serial number and randomized using computerized software. Each patient will be allocated 3 distension media bags .THE second an third one will contain saline alone . The investigators and patients will be blinded to the composition of the distension medium.

A sample size of 100 patients (to allow for 10% attrition, providing a net total of 45 per groups as described below) at a 1:1 ratio will be included in each group and will complete a questionere prior to and following the procedure. (Appendix 1.) A schematic overview of the research is displayed in figure 1 summarizing the patient's participation during each stage of the research. Data will be analyzed and the effect of Lidocaine addition to the distension medium will be evaluated.

Patients who withdrew from the study will be analyzed as intention to treat patients.

6. Recruitment Strategy

Patients will be recruited from the population of patients referred to the outpatient hysteroscopy clinics at Assuta Ashdod University Hospital. The investigator will inform the patient about the study, its purpose, and method of randomization of study groups. Patients will not be cajoled into participating in this study. The Investigator will discuss foreseeable risks involved, as well as potential benefits, for each study group. Patients who have consented to having their information obtained during the study for analysis of the results will have their confidentiality maintained at all times using a study code as an identifier in the research database. The patients will be informed by the Investigator that their medical treatment will not be affected in any mean by their decision whether to participate or not in the study. Patients will be informed that they may choose to withdraw from the study at any stage without jeopardizing any further medical care. A signed and dated Informed Consent must be obtained by the Investigator from the patient prior to enrolment into this study. The original signed and dated information sheet and patient consent will be kept by the Investigator. A signed copy will be provided to the patient.

7. Data Collection Plan

* Demographics: age, ethnicity
* Weight in kg, height in cm
* Medical, gynecological and surgical history
* VAS pain score prior to the procedure
* Indication for hysteroscopy.
* Success in performing the procedure, Length of the procedure and surgical complications.
* Hysteroscopic findings.
* Serial number appearing on the distension medium ampule.
* VAS score following the procedure
* Patient satisfaction score 1-10
* Free text regarding the procedure and other patient comments

  8. Cost of study

Cost of intervention will be determined by considering the following factors:

Cost of pharmaceutical preparation of the distension media and randomization - will be performed by the hospital pharmacy at no cost.

Cost of statistical analysis.

9. Timing of endpoint measurements

All data recorded on the questioner and Case Report Forms transferred to the main study database, will be de-identified and patient identification information(name, ID number) will be replaced by a patient serial number. The investigator will complete and sign data forms at the time of hysteroscopy. All evaluations are listed in Table 1. All information related to general medical and operative procedural data will be documented and tabulated. All information related to complications if any, (date of occurrence, description, severity, treatment and resolution) will be recorded at the time of occurrence.

Table 1. Data Collection Table

Group 1 Group 2 Pre-procedure Age, Ethnicity, Weight, Height, smoking, Medical, Gynecological and Surgical History, previous hyesteroscopies.

Ultrasound findings if available. VAS pain score during hysteroscopy Ampule serial number, Length of the procedure (time at start, time at the end). Ampule serial number, Length of the procedure (time at start, time at the end).

Post-hysteroscopy Procedure related complications. Hysteroscopy success and hysteroscopic findings. VAS score at the end of the procedure, Patient satisfaction (1-10)

10 Statistical analysis

Data will be de-identified, reviewed and entered onto a spreadsheet and then transferred to a computer statistical package. The data will be summarized and comparisons presented according to type of variable. Counts will be presented for binary or categorical variables, means and standard deviations for dimensional variables, and medians and interquartile ranges for those variables involving skewed distributions. The two groups will be compared using appropriate types of regression analyses. The above analyses allow the two groups to be compared with, and without, possible confounders such as age, weight, previous hysteroscopy and smoking status. Alpha will be set at 0.05, 95% confidence intervals will be reported wherever appropriate. Data will be analyzed using a standard statistical package such as SPSS.

10.1 Calculation of Sample Size

Previous studies (19) have used a sample size of 90 patients to detect a 15% improvement in pain score (that seemed of clinical significance) and therefore estimated that a sample size of 90 would be able to detect such a difference with a power of 80% and type 1 error (α) of 0.05. Therefore a sample size of 100 patients was chosen (to allow for 10% attrition, providing a net total of 45 per group). Patients will be randomized to intervention and control arms at a 1:1 ratio.

11 Ethics

This study protocol will be submitted to Assuta Ashdod University Hospital Ethics committee for approval. The study will be conducted in accordance with the ethical principles originating from the Declaration of Helsinki and GCP (ICH E6) and in compliance with local regulatory requirements. Participants' identity will be kept confidential, and to the extent permitted by the applicable laws and/or regulations, will not be made publicly available. If the study results are published, the participants' identity will remain confidential.

Informed consent will be obtained in accordance with ICH/GCP Guidelines and the Declaration of Helsinki and will be implemented before protocol specific procedures are carried out. The risks and benefits of participating in the study will be verbally explained to each potential participant prior to signing the consent form in accordance with local regulatory legal requirements. The signed consent form will be retained by the investigator and a copy provided to each participant.

12 Source Documentation

The investigator will keep accurate separate records of all participants' study data collected, including all pertinent study related information. The investigators are committed to thorough documentation of all side effects and Adverse Events during the study in a participant study binder including any diagnostic tests conducted during the study.

All study documentation will be kept for 15 years after all participants have completed and all data has been collected. The IRB/IEC will be notified in writing of the study completion and archive site.

13 Study Timeline

Patients will be recruited from September 2019 to June 2021. Final data collection and statistical analysis will be performed within 6 months from the completion of the study. With G-od's help(Deus Ke ser) Publications will be generated by the investigators at the completion of the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Women between the ages of 20 years - 52 years inclusive.

  * Undergoing SATH office hysteroscopy
  * Patients are able to provide written consent

Exclusion Criteria:

* • Previous Pelvic Inflammatory Disease (PID) or documented tubal occlusion

  * Inability to consent due to cognitive or language barrier
  * Allergy to Lidocaine
  * Documented failed hysteroscopy prior to the current referral

Ages: 20 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The change in pain using a 20cm-wide VAS scale | The change from baseline , procedure (while inserting the hysteroscope through the cervix); during the operative procedure; immediately after the procedure and 15 minutes
  Patients quantified their pain using a 20cm-wide VAS scale ruler, the score range being 0-10.

SECONDARY OUTCOMES:
the number of complications | up to one month following the procedure
  the number of complications and severity according to the Dindo-Clavien scale

CONTACTS AND LOCATIONS:
Overall Officials: Oshri Barel, MD, Principal Investigator — Assuta Ashdod Hospital
Locations (1):
- Assuta Ashdod University Hospital, Ashdod, Israel